CLINICAL TRIAL: NCT06308705
Title: The SsRI/NIE Recombinant Antigen ELISA for the Follow up of Patients Infected by Strongyloides Stercoralis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-19
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Strongyloides Stercoralis Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sera (Other): All sera available in our biobank and originating from the Strong Treat trial will be eligible for the study, based on the availability of the baseline and the 12-month follow up serum of each included case.
  Interventions: Diagnostic Test: InBios Strongy Detect TM IgG ELISA

INTERVENTIONS:
Diagnostic Test: InBios Strongy Detect TM IgG ELISA — The InBios Strongy Detect TM IgG ELISA detects specific IgG antibodies to Strongyloides recombinant antigens NIE and SsIR in serum. It consists of an enzymatically amplified sandwich-type immunoassay. Positive and negative control samples are provided in the kit. The test will be run and interpreted according to the manufacturer's instruction. The results are expressed as OD and nOD. Clinical interpretation of the results will be done by analysis of the Receiver Operating Characteristics (ROC) curve generated using data from confirmed positive and confirmed negative samples.

SUMMARY:
This is a single-center interventional study with an IVD medical device.

The main objective of this study is to evaluate the ELISA SsIR/NIE test for the post-treatment follow-up of patients suffering from strongyloidosis, using well-characterized sera from a previous study.

All sera available in the Tropica biobank and coming from the Strong Treat study, for which serum samples collected at baseline and at 12-month follow-up are available, will be eligible for the study.

The test The InBios Strongy Detect TM IgG ELISA detects specific IgG antibodies against recombinant Strongyloides NIE and SsIR antigens in serum. It consists of an enzymatically amplified sandwich immunoassay. Positive and negative control samples are provided in the kit. The test will be performed and interpreted according to the manufacturer's instructions. The results are expressed as OD and nOD. Clinical interpretation of the results will be performed by receiver operating characteristic (ROC) curve analysis generated using data from confirmed positive and confirmed negative samples.

The laboratory technicians will receive from the PI of the study a list of pseudo-anonymized sera to be tested with SsIR/NIE ELISA, they will check their availability and proceed with the test according to the Manufacturer's instructions. Laboratory personnel performing and reading the tests will be blinded to the results of any previously performed tests (and the classification of the sample in the Strong Treat study). A single run will be performed for each sample, unless the test needs to be repeated due to any technical problem. Both baseline and follow-up sera will be tested. The resulting OD and nOD will be reported in an Excel file by the laboratory technicians performing the tests.

ELIGIBILITY:
Inclusion Criteria:

* All sera available in our biobank and originating from the Strong Treat trial
* availability of the baseline and the 12-month follow up serum of each included case

Exclusion Criteria:

* unavailability of the baseline or of the 12-month follow up serum of each included case

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Result of the SsIR/NIE ELISA | Baseline and at the 12-month follow-up
  For each sample, the result of the SsIR/NIE ELISA will be compared with the outcome category (cure/persistence of infection) defined at the 12-month follow up within the Strong Treat study. Similarly to what is established with other serology tests, SsIR/NIE ELISA will indicate parasitological cure when at least a twofold reduction of nOD at the 12-month follow up, compared to the baseline nOD, will be observed.

SECONDARY OUTCOMES:
Seroconversion | Baseline and at the 12-month follow-up
  Proportion of SsIR/NIE ELISA tests showing complete seroreversion within the subgroup of cases that will be correctly (in comparison with the Strong Treat category) classified as cured by the SsIR/NIE ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy